CLINICAL TRIAL: NCT04572880
Title: Evaluation of Minimal Invasive Glaucoma Surgery: Trabeculectomy vs. XEN ® vs. Preserflo ®. Randomized Clinial Trial
Brief Title: Evaluation of Minimal Invasive Glaucoma Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Lindner Ewald, MD, Priv.-Doz. Dr.med.univ. Lindner Ewald, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1234567
Record Dates: First submitted 2020-08-03; First posted 2020-10-01 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Glaucoma
Keywords: MIGS; XEN®; Trabeculectomy; Preserflo®
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Trabeculectomy (Active Comparator)
  Interventions: Procedure: Trabeculectomy
- XEN® (Active Comparator)
  Interventions: Device: XEN®
- Preserflo® (Active Comparator)
  Interventions: Device: Preserflo®

INTERVENTIONS:
Procedure: Trabeculectomy — Trabeculectomy is performed
  Arms: Trabeculectomy
Device: XEN® — Microinvasive Surgery with XEN® is performed
  Arms: XEN®
Device: Preserflo® — Microinvasive Surgery with Preserflo® is performed
  Arms: Preserflo®

SUMMARY:
Glaucoma is a neurodegenerative disease with an accelerated and progressiv retinal ganglion cell loss and concomitant visual field defects. Glaucoma can be treated with eye drops, laser therapy or surgery. Various surgical approaches to lower intraocular pressure are available, amongst which trabeculectomy is the gold standard. Recently minimal invasive glaucoma surgery has been introduced and has become a good alternative to trabeculectomy. Randomized clinical trials investigating the postoperative outcomes of various types of glaucoma surgery are limited.

DETAILED DESCRIPTION:
150 Patients will be randomized to one of the 3 surgeries. Trabeculectomy Preserflo® or Xen® will be done according to a standard protocol Data will be collected for 5 years after surgery, Visual Acuity, Applanation Tonometry, Slit lamp Biomicroscopy, Endothelial cell cound, visual fields, optical coherence tomography of the optic disc, retina and anterior segment, impression cytology and life quality will be done on day of enrollment and during followup. Mean Intraocular pressure and number of glaucoma medications, Endothelial cell loss, visual acuity, visual fields and assessment of life quality will be assessed during the post-operative follow-ups at one week, one month, 3 months, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patiens with glaucoma in which surgery is indicated to reach target intraocular pressure
* Subjects not anticipated to require any further surgery in the next 12 months

Exclusion Criteria:

* Patients who do not want to make follow-ups at the department
* angle closure, uveitic, neovascular, congenital glaucoma, iridocorneal endothelial syndrom, Axenfeld-Rieger syndrom.
* Prior filtering glaucoma surgery, suprachoroidal stent, retinal surgery, corneal graft surgery or cyclophotocoagulation
* Any major ocular inflammation up to 30 days prior to surgery
* Conjunctival scarring
* Allergy to any drugs required for the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Mean intraocular pressure | up to 5 years post surgery
  Goldmann Applanation Tonometry [mmHg]

SECONDARY OUTCOMES:
Number of medications | up to 5 years post surgery
  antihypertensive eye-drops

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria